CLINICAL TRIAL: NCT06285942
Title: EdOxaban in fRagIle Patients With Percutaneous Endoscopic GAstrostoMy and atrIal fIbrIllation: the ORIGAMI II Study
Brief Title: EdOxaban in fRagIle Patients With Percutaneous Endoscopic GAstrostoMy and atrIal fIbrIllation
Acronym: ORIGAMI II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Domenico D'Amario, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 277.535; CE366/2023 (Registry Identifier: CET AOU Maggiore della Carità di Novara)
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Fragility
Keywords: Edoxaban; Fragile Patient; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An interim-analysis will be performed on the primary endpoint when at least 50% of patients will have been randomized and completed the 6 months follow-up. The interim-analysis will be performed by an independent statistician, blinded for the treatment allocation. The statistician will report to the independent data and safety monitoring board
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Edoxaban (Experimental): This arm will receive Edoxaban via PEG
  Interventions: Drug: Edoxaban
- No Edoxaban (Active Comparator): This arm will receive other DOACs through PEG or subcutaneous heparin or LMWH
  Interventions: Drug: No Edoxaban

INTERVENTIONS:
Drug: Edoxaban — To use of Edoxaban via PEG in patients with an indication to anticoagulation therapy according to current guidelines
  Arms: Edoxaban
Drug: No Edoxaban — Other DOACs through PEG or subcutaneous heparin or LMWH
  Arms: No Edoxaban

SUMMARY:
The goal of this interventional study is to describe the use of Edoxaban via PEG in patients with an indication to anticoagulation therapy. One arm will receive Edoxaban through PEG and the other arm will receive other Direct oral anticoagulants through PEG or subcutaneous heparin or LMWH.

Once enrolled, patients will be treated with a single daily dose of Edoxaban (60 or 30 mg according to specific indications). At day 4 after enrollment (steady state), evaluation of anti-FXa activity and thrombin generation assay will be performed on peripheral whole blood samples. At months 6 and 12 patients will be asked to complete the ACTS (Anti-Clot treatment scale) questionnaire specific for anticoagulation.

The main endpoint will be: the difference in the results of the Anti-Clot treatment scale questionnaire between the two groups evaluated at 12 months.

DETAILED DESCRIPTION:
Direct oral anticoagulants (DOAC) have a remarkable efficacy/safety ratio, a predictable anticoagulant effect and are recommended by ESC guidelines to be preferred over vitamin K antagonist (VKA) wherever possible in the prevention of stroke and systemic embolism in adult patients with non-valvular atrial fibrillation. Enteral access feeding devices are placed in patients who have a functional and accessible gastrointestinal tract but are not able to maintain an adequate oral intake. Among these devices, percutaneous endoscopic gastrostomy (PEG) represents a valid option, especially for long-term feeding, and PEG positioning has shown a steadily increasing trend in fragile patients with several comorbidities.

A significant subgroup of subjects with PEG tube has an indication to long-term anticoagulant therapy, mainly represented by atrial fibrillation. Among the several pharmacodynamic pathway mediating anticoagulation, direct FXa inhibitors block both free FXa and FXa bound to form the prothrombinase complex, whereas the indirect FXa inhibitors, such as LMHW, only inhibit free FXa. It was recently described a safe and effective anticoagulation through the administration of edoxaban 30 mg daily (crushed and diluted in 10 mL of saline solution) through a PEG in a patient with advanced amyotrophic lateral sclerosis, tracheostomy, atrial fibrillation, and a recent acute heart failure. On these premises, the investigators designed the ORal anti-coagulants In fraGile patients with percutAneous endoscopic gastrostoMy and atrIal fibrillation (ORIGAMI) pilot investigation, evaluating the feasibility, anticoagulant effectiveness and preliminary safety and efficacy of edoxaban administration via PEG in fragile patients with NVAF requiring long-term anticoagulation treatment.

The ORIGAMI II study will be a prospective, multi-centre, double arm, open label, clinical trial, aiming to describe the use of Edoxaban via PEG in patients with an indication to anticoagulation therapy according to current guidelines. One arm will receive Edoxaban through PEG and the other arm will receive other DOACs through PEG or subcutaneous heparin or LMWH.

The study will enroll 168 patients, who will be followed-up for 12 months. The Centers that will participate in this study will be: the AOU Maggiore della Carità of Novara (as coordinating center); Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma; Ospedale Policlinico San Martino, Genova.

The primary endpoint of this study is the difference in Anti-Clot treatment scale questionnaire results among the two groups assessed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PEG (recent implantation or already present)
* Indication for long-term oral anticoagulation

Exclusion Criteria:

* Under 18 years of age
* Life expectancy <30 days
* Lack of informed consent
* Contraindication to DOACs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Anti-Clot treatment scale (ACTS) questionnaire results among the two groups assessed at 6 and 12 months. | at 6 and 12 months
  The Anti-Clot treatment scale (ACTS) is a 15-item patient-reported instrument of satisfaction with anticoagulant treatment. It includes a 12-item ACTS Burdens scale and a 3-item ACTS Benefits scale. The rate of experience of anticoagulant treatment during the past 4 weeks on a 5-point scale of intensity: 1 = not at all, 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely.

SECONDARY OUTCOMES:
Number of cardio-embolic events at 6 and12 months | at 6 and 12 months
  The number of cardio-embolic events consisting of stroke, systemic embolism or symptomatic relapse of deep vein thrombosis/pulmonary embolism.
Number of bleeding events | at 6 and 12 months
  The Bleeding Academic Research Consortium (BARC) scale and the Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria will be considered.
  BARC scale from Type 1 (bleeding that is not actionable) to Type 5b (Fatal bleeding); TIMI bleeding criteria range from Minimal to Major, such as any intracranial bleeding, clinically evident signs of hemorrhage associated with a drop in hemoglobin ≥ 5 g/dl or fatal bleeding.
Assessment of drugs efficacy by measuring the anti-factor Xa activity | at 6 and 12 months
  Mean DOACs plasma concentration-time profile will be measured at steady state as anti-FXa activity using the STA®-Liquid Anti-Xa assays on a STA Compact Max® instrument. The evaluation of the anti-FXa activity will be performed on peripheral whole blood samples.
Assessment of drugs efficacy by measuring the thrombin generation | at 6 and 12 months
  At steady state will be measured the thrombin generation assay, both in patients receiving DOACs and in those receiving parenteral anticoagulation. The evaluation of the thrombin generation assay will be performed on peripheral whole blood samples.
Assess the quality of life | at 6 and 12 months
  The Zarit Burden Interview (ZBI) will be used to assess quality of life. The ZBI is an interview to evaluate the consequences that the care burden of a family member with chronic or degenerative pathologies has on the caregiver, with a scale ranging from 0 with zero care load, to 88 with a maximum level of care load.
Cost-effectiveness analysis | at 6 and 12 months
  A cost-effectiveness analysis will be carried out to compare the costs (direct and indirect) of treatment with Edoxaban compared to other subcutaneous anticoagulants.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale Policlinico San Martino, Genova
  - AOU Maggiore della Carità, Novara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galli M, Andreotti F, Porto I, Crea F. Intracranial haemorrhages vs. stent thromboses with direct oral anticoagulant plus single antiplatelet agent or triple antithrombotic therapy: a meta-analysis of randomized trials in atrial fibrillation and percutaneous coronary intervention/acute coronary syndrome patients. Europace. 2020 Apr 1;22(4):538-546. doi: 10.1093/europace/euz345. PMID 31942971
- [Background] Galli M, Porto I, Andreotti F, D'Amario D, Vergallo R, Della Bona R, Crea F. Early anticoagulation in the current management of NSTE-ACS: Evidence, guidelines, practice and perspectives. Int J Cardiol. 2019 Jan 15;275:39-45. doi: 10.1016/j.ijcard.2018.10.087. Epub 2018 Oct 27. PMID 30391063
- [Background] Galli M, D'Amario D, Andreotti F, Porto I, Vergallo R, Sabatelli M, Lancellotti S, Meleo E, De Cristofaro R, Crea F. Sustained safe and effective anticoagulation using Edoxaban via percutaneous endoscopic gastrostomy. ESC Heart Fail. 2019 Aug;6(4):884-888. doi: 10.1002/ehf2.12434. Epub 2019 Jun 11. PMID 31184800
- [Background] D'Amario D, Galli M, Canonico F, Restivo A, Arcudi A, Scacciavillani R, Cappannoli L, Riccioni ME, Annetta MG, Di Stefano G, Piccinni C, Vergallo R, Montone RA, Leone AM, Niccoli G, Sabatelli M, Antonelli M, Andreotti F, De Cristofaro R, Crea F. ORal anticoagulants In fraGile patients with percutAneous endoscopic gastrostoMy and atrIal fibrillation: the (ORIGAMI) study. J Cardiovasc Med (Hagerstown). 2021 Mar 1;22(3):175-179. doi: 10.2459/JCM.0000000000001142. PMID 33186237
- [Background] D'Amario D, Galli M, Cappannoli L, Canonico F, Restivo A, Arcudi A, Scacciavillani R, Riccioni ME, Vergallo R, Montone RA, Conte A, Meleo E, Lancellotti S, Sacco M, Antonelli M, Andreotti F, DE Cristofaro R, Crea F. Oral anticoagulants in fragile patients with percutaneous endoscopic gastrostomy and atrial fibrillation: the ORIGAMI pilot investigation. Minerva Cardiol Angiol. 2023 Feb;71(1):109-116. doi: 10.23736/S2724-5683.21.05903-2. Epub 2022 Feb 15. PMID 35166091